CLINICAL TRIAL: NCT03950973
Title: Improving Diabetes Outcomes and Health Disparities Through a Patient Activation Intervention Addressing Unmet Resource Needs
Brief Title: Diabetes Outcomes and Unmet Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Minal Patel, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUM00149794; R01DK116715 (NIH)
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetes
Keywords: Diabetes; Self-management; Adherence; Social determinants of health; Social risk factors
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CareAvenue (Experimental): Participants receive access to CareAvenue, an e-health tool, and receive one weekly automated telephone call and 4-5 text messages per week for 52 weeks.
  Interventions: Behavioral: CareAvenue
- Guest Assistance Program (Active Comparator): Participants receive information about the Guest Assistance Program (GAP) and receive 3-4 text messages per week related to diabetes management and resources for 52 weeks.
  Interventions: Behavioral: Guest Assistance Program

INTERVENTIONS:
Behavioral: CareAvenue — CareAvenue is an e-health tool providing information about diabetes management and low-cost resources. Participants in this group have access to CareAvenue and receive a weekly automated phone call and text messages related to CareAvenue and its resources as well as diabetes management.
  Arms: CareAvenue
Behavioral: Guest Assistance Program — The Guest Assistance Program (GAP) is a resource, which provides assistance with medical and non-medical needs and resources to patients receiving medical care at University of Michigan health system. Participants in this group are provided with GAP information and receive text messages related to diabetes management.
  Arms: Guest Assistance Program

SUMMARY:
This study will refine and test the effectiveness of CareAvenue, an automated e-health tool that informs and activates patients with uncontrolled diabetes to take steps in accessing resources and engaging in self-care. Our central hypothesis is that activating patients with uncontrolled diabetes and linking them to resources to address financial burden and unmet social risk factors will improve both intermediate outcomes and measures of disease control above and beyond existing services, especially for high need patients.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-75 years of age
* Be diagnosed with type 1 or type 2 diabetes with prescribed anti-hyperglycemic medication
* Have a most recent hemoglobin A1c(HbA1c) level within the past 6 months of ≥7.5% for individuals ≤70 years and >8.0% for individuals between 70-75 years in age
* Have access to a telephone that can receive and send text messages
* Not participating in another diabetes intervention research study

Exclusion Criteria:

* Significant cognitive impairment precluding individuals from completing the study as evidenced by ability to complete study intake procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minal R Patel, PhD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underlie results in a publication, after de-identification.
Supporting Information: SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: The data will be made available to other researchers who provide a methodologically sound proposal and who have appropriate approvals from all relevant IRBs. The data will be shared for analyses to achieve aims in the approved proposal. Data will be shared through a secure FTP site through encryption protocols that allow secure uploading of files with data sharing limited to specific users. Select datasets will also be made available through the University of Michigan openICPSR Repository (http://www.icpsr.umich.edu/icpsrweb/deposit/index.jsp). Proposals should be directed to minalrp@umich.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Patel MR, Zhang G, Heisler M, Piette JD, Resnicow K, Choe HM, Shi X, Song P. A Randomized Controlled Trial to Improve Unmet Social Needs and Clinical Outcomes Among Adults with Diabetes. J Gen Intern Med. 2024 Oct;39(13):2415-2424. doi: 10.1007/s11606-024-08708-8. Epub 2024 Mar 11. PMID 38467918
- [Derived] Patel MR, Heisler M, Piette JD, Resnicow K, Song PXK, Choe HM, Shi X, Tobi J, Smith A. Study protocol: CareAvenue program to improve unmet social risk factors and diabetes outcomes- A randomized controlled trial. Contemp Clin Trials. 2020 Feb;89:105933. doi: 10.1016/j.cct.2020.105933. Epub 2020 Jan 7. PMID 31923472

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening eligible and consenting to participate, 67 participants either later changed their mind and declined to participate prior to starting data collection, were unreachable for baseline collection, or did not complete baseline in order to be randomized.
Groups:
- CareAvenue (Intervention): Participants receive access to CareAvenue, an e-health tool, and receive one weekly automated telephone call and 4-5 text messages per week for 52 weeks.
  CareAvenue: CareAvenue is an e-health tool providing information about diabetes management and low-cost resources. Participants in this group have access to CareAvenue and receive a weekly automated phone call and text messages related to CareAvenue and its resources as well as diabetes management.
- Guest Assistance Program (Control): Participants receive information about the Guest Assistance Program (GAP) and receive 3-4 text messages per week related to diabetes management and resources for 52 weeks.
  Guest Assistance Program: The Guest Assistance Program (GAP) is a resource, which provides assistance with medical and non-medical needs and resources to patients receiving medical care at University of Michigan health system. Participants in this group are provided with GAP information and receive text messages related to diabetes management.
Period: Overall Study
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Started | 301 (Allocated to Intervention) | 299 (Allocated to Control)
Follow Up 1 Completion (Completed next data collection timepoint (Follow-Up 1)) | 206 (Completed next data collection timepoint (Follow-Up 1)) | 258 (Completed next data collection timepoint (Follow-Up 1))
Follow Up 2 Completion (Completed final data collection timepoint (Follow-Up 2)) | 196 (Completed final data collection timepoint (Follow-Up 2)) | 239 (Completed final data collection timepoint (Follow-Up 2))
Completed | 196 (Completed final data collection timepoint (Follow-Up 2)) | 239 (Completed final data collection timepoint (Follow-Up 2))
Not Completed | 105 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control) | Total
Number analyzed (Participants) | 301 | 299 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.64 (13.68) | 54.26 (12.33) | 53.45 (1304)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 168 | 166 | 334
  Gender: Male | 132 | 132 | 264
  Gender: Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Several participants refused to answer survey questions on race and ethnicity
  Participants
    Race: number analyzed (Participants) | 300 | 298 | 598
    Race: Non-Hispanic White | 204 | 184 | 388
    Race: Non-Hispanic Black | 43 | 58 | 101
    Race: Hispanic | 16 | 15 | 31
    Race: Asian | 9 | 14 | 23
    Race: Multiple Race | 22 | 20 | 42
    Race: Other | 6 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 301 | 299 | 600
Income as percent of poverty level [Count of Participants; unit: Participants] — Population: Several participants refused to answer survey question about income
  Participants
    number analyzed (Participants) | 297 | 296 | 593
    Less than 100% | 35 | 38 | 73
    100-200% | 52 | 43 | 95
    201-400% | 131 | 130 | 261
    Greater than 400% | 79 | 85 | 164
Type of diabetes [Count of Participants; unit: Participants]
  Type 1 | 61 | 69 | 130
  Type 2 | 240 | 230 | 470
Number of chronic conditions [Mean (Standard Deviation); unit: number of chronic conditions] | 4.12 (2.31) | 4.18 (2.31) | 4.15 (2.31)
Health Insurance Type [Count of Participants; unit: Participants]
  None | 2 | 9 | 11
  Private | 132 | 128 | 260
  Medicare | 19 | 25 | 44
  Medicaid | 45 | 34 | 79
  Medicare + Medicaid Supplemental | 34 | 30 | 64
  Medicare + Private Supplemental | 68 | 72 | 140
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c as Measured by an HbA1c Machine
Description: HbA1c will be measured at baseline, 6 months, and 12 months using HbA1c machine. HbA1c is a measure of the average level of glucose in blood over the past 3 months measured as a percentage.
  The change in HbA1c from baseline to 12 months is reported here as the primary outcome.
Time Frame: Assessed at Baseline, 6 months, 12 months (Change between baseline and 12 months reported)
Population: Change from baseline to 12-month follow-up The overall number of participants analyzed is different from the participant flow module due to missingness, unable to obtain measurement, etc.
Measure: Mean (Standard Deviation); unit: percentage of average glucose 3 months
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Number analyzed (Participants) | 193 | 233
percentage of average glucose 3 months | 0.07 (1.57) | -0.10 (1.42)

2. Secondary Outcome: Change in Systolic Blood Pressure as Measured an Automated Blood Pressure Machine
Description: Systolic blood pressure will be measured at baseline, 6 months, and 12 months using an automated blood pressure machine in millimeters of mercury (e.g., 120 mm Hg).
  The change in systolic blood pressure from baseline to 12 months is reported here as secondary outcome.
Time Frame: Assessed at Baseline, 6 months, 12 months (Change between baseline and 12 months reported)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Number analyzed (Participants) | 193 | 239
mmHg | -4.00 (18.83) | -6.00 (19.92)

3. Secondary Outcome: Change in Cost-Related Non-Adherence Behaviors With Prescribed Treatment Regimens Related to Diabetes as Measured by Participant Questionnaire
Description: Cost-Related Non-Adherence (CRN) Behaviors related to diabetes will be measured at baseline, 6 months, and 12 months by 4-items adapted from the Medicare Current Beneficiary Survey and 2 items adapted from the National Health Interview Survey that look at diabetes. The items are measured with a 4-point Likert scale. Participants answering "often" or "sometimes" to any of the items are indicated as exhibiting CRN. Min value of 0, max value of 18, with higher scores indicating more cost-related non-adherence behaviors.
  The change in CRN behaviors from baseline to 12 months is reported here as the secondary outcome.
Time Frame: Assessed at Baseline, 6 months, 12 months (Change between baseline and 12 months reported)
Population: Change from baseline to 12-month follow-up The overall number of participants analyzed is different from the participant flow module due to missingness
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Number analyzed (Participants) | 196 | 238
score on a scale | -0.45 (3.52) | -0.91 (3.62)

4. Secondary Outcome: Change in Cost-Related Non-Adherence Behaviors With Prescribed Treatment Regimens Related to Other Conditions Being Managed as Measured by Participant Questionnaire
Description: Cost-Related Non-Adherence (CRN) Behaviors related to other conditions being managed will be measured at baseline, 6 months, and 12 months by 4-items adapted from the Medicare Current Beneficiary Survey and 2 items adapted from the National Health Interview Survey that look at other health conditions being managed. The items are measured with a 4-point Likert scale. Participants answering "often" or "sometimes" to any of the items are indicated as exhibiting CRN. Mean values were obtained, with min value of 0, max value of 1, with higher mean scores indicating more cost-related non-adherence behaviors.
  The change in CRN behaviors from baseline to 12 months is reported here as the secondary outcome.
Time Frame: Assessed at Baseline, 6 months, 12 months (Change between baseline and 12 months reported)
Population: Change from baseline to 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Number analyzed (Participants) | 196 | 239
score on a scale | -0.07 (0.45) | -0.06 (0.48)

5. Secondary Outcome: Change in Perceived Financial Burden as Measured by the Comprehensive Score for Financial Toxicity (COST) - Functional Assessment of Chronic Illness Therapy (FACIT)
Description: Perceived Financial Burden will be measured at baseline, 6 months, and 12 months by the 11-item measure Comprehensive Score for Financial Toxicity (COST) - Functional Assessment of Chronic Illness Therapy (FACIT) that were measured on a 5-point scale (0: not at all - 4: very much). The score includes reverse-coding 6-items, summing all items, multiplying sum by 11 and dividing the total by number of items answered. Lower scores indicate higher perceptions of financial burden. (Min value of 0, max value of 44) The change in perceived financial burden (COST measure) from baseline to 12 months is reported here as secondary outcome.
Time Frame: Assessed at Baseline, 6 months, 12 months (Change between baseline and 12 months reported)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Number analyzed (Participants) | 195 | 238
score on a scale | 2.01 (7.47) | 2.74 (7.36)

6. Secondary Outcome: Change in Unmet Social Risk Factors as Measured by 20 Items in Participant Questionnaire
Description: Change in Unmet Social Risk Factors will be measured at baseline, 6 months, and 12 months by 20 items adapted from the Accountable Health Communities Health-Related Social Needs Screening Tool, the Health Leads Social Needs Screening Toolkit, and the Kaiser Permanente Your Current Life Situation Questionnaire. The item values are binary (yes/no). Higher number of "yes" responses indicates higher number of unmet social risk factors/higher need. (Min value of 0, max value of 20).
  The change in unmet social risk factors from baseline to 12 months is reported here as secondary outcome.
Time Frame: Assessed at Baseline, 6 months, 12 months (Change between baseline and 12 months reported)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: yes responses
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Number analyzed (Participants) | 195 | 238
yes responses | -1.05 (3.69) | -1.48 (4.10)

7. Secondary Outcome: Change in Unmet Social Risk Factors as Measured by Participant Questionnaire
Description: Change in Unmet Social Risk Factors will be measured at baseline, 6 months, and 12 months by 3 items from the Accountable Health Communities Health-Related Social Needs Screening Tool and 1 item adapted from the National Health Interview Survey. The items each have three response options, in which a positive response indicates an unmet social risk factor. Higher scores indicate more unmet social risk factors (min value of 0; max value of 8).
  The change in unmet social risk factors from baseline to 12 months is reported here as secondary outcome.
Time Frame: Assessed at Baseline, 6 months, 12 months (Change between baseline and 12 months reported)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
Number analyzed (Participants) | 194 | 238
units on a scale | -0.26 (1.42) | -0.27 (1.38)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 1 year time period (from completing study consent to completing final data collection).
Description: Adverse Events were monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated
Arm/Group | CareAvenue (Intervention) | Guest Assistance Program (Control)
All-Cause Mortality (participants affected / at risk) | 2/301 | 2/299
Serious Adverse Events (participants affected / at risk) | 123/301 | 125/299
Other Adverse Events (participants affected / at risk) | 75/301 | 86/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CareAvenue (Intervention) (N=301) | Guest Assistance Program (Control) (N=299)
Hospitalization (Infections and infestations) | 15 (19) | 10 (11)
Hospitalization (Surgical and medical procedures) | 12 (13) | 12 (13)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) | 2 (3) — Blood Pressure
Hospitalization (Metabolism and nutrition disorders) | 4 (4) | 6 (6) — Blood sugar
Hospitalization (General disorders) | 10 (12) | 15 (18) — Organ System related or Other
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) — COVID
Death (General disorders) | 2 (2) | 2 (2)
Other Serious Event (General disorders) | 87 (112) | 99 (140)
Hospitalization (General disorders) | 9 (11) | 15 (17) — Other
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CareAvenue (Intervention) (N=301) | Guest Assistance Program (Control) (N=299)
Other Non-Serious Adverse Events (General disorders) | 75 (110) | 86 (105) — Includes unexpected/unrelated, expected/unrelated, expected/related, and unexpected/related (all non-serious) adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03950973/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03950973/ICF_001.pdf